CLINICAL TRIAL: NCT04267458
Title: the Prevalence of Acute Kidney Injury in Patients With Chronic Hepatitis c Virus Receiving Sofuspovir Containing Direct Acting Antiviral Therapy
Brief Title: Prevalence of Kidney Injury in Patients With HCV Treated With Sofuspovir Containing DAA Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia K. Zaafar, lecturer of pharmacology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-2019
Record Dates: First submitted 2020-01-26; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Investigate the Renal Effect of DAAs on Egyption Patients After Completion of Treatment
Keywords: DAA; HCV; egyption patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCV infected patients with non-elevated sCr than basal levels (Other): a group of egyption patients with HCV infection with non-elevated sCr than basal levels and treated with sofuspovir as an direct acting antiviral drug
  Interventions: Other: evaluation of sofuspovir containing DAA regien expected insult on kidney

INTERVENTIONS:
Other: evaluation of sofuspovir containing DAA regien expected insult on kidney — to use different kidney biomarkers to evaluate acute kidney damage after using sofuspovir containing DAA regimen in treatment of HCV

SUMMARY:
this study aims is to investigate the occurrence of AKI during antiviral therapy, defined as an increase of 0.3 mg/dL or 50% at least in serum creatinine level when compared with baseline values or more than a 25% reduction in (eGFR) when compared with baseline eGFR in Egyptian patients.In addition to evaluate the change in insulin resistance value after treating patients from HCV.

DETAILED DESCRIPTION:
There are limited published data, currently, suggesting the risk of AKI during oral direct acting antiviral treatment. Most case reports and retrospective studies reported the presence of an intrinsic cause of renal injury, with most of the available biopsies showing acute tubular necrosis (ATN) and acute interstitial nephritis (AIN). Most of these patients had returned to baseline renal function on cessation of sofosbuvir combination therapy.

Recently it was found that a notable percentage of patients experienced a transient increase in creatinine during therapy, which could occasionally lead to a more than 50% decrease in patients' eGFR. Previous studies had also shown that the co-use of nonsteroidal anti-inflammatory drugs (NSAIDs) and recurrent ascites were at increased risk for AKI during sofosbuvir-based antiviral therapy.

The primary endpoint of this study is to investigate the occurrence of AKI in Egyptian patients during antiviral therapy and to highlight its reasons and time of incidence in addition to the mechanism of this injury.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from HCV
* male or female
* easy to treat naive patients

Exclusion Criteria:

* pregnant women
* seffering from HBV
* diffecult to treat
* other comorbodities as heart diseases or COPD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
investigate the renal injury which can be caused during using sofuspovir containing DAA regimen in HCV treatment | from the start to 6 months later
  to investigate effect of DAA on kidney of treated patients and the mechanism of the drug to cause this renal effect by causing renal buimarkers including NAG and eGFR

SECONDARY OUTCOMES:
highlight the effect of DAAs on insulin resistance in diabetic patients suffering from HCV | from the starting of treatment till the 3-months follow up after the end of the treatment regimen
  to estimate the effect of DAAs on HOMA-IR index f insulin resistance in diabetic infected patients and comparing their insulin resistance before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Zaafar, PhD, Principal Investigator — Lecturer of pharmacology and toxicology
Locations (1):
- Thabet Thabet Hospital For Internal Diseases, Cairo, Egypt